CLINICAL TRIAL: NCT00703521
Title: A Three-Year Clinical Study on Immunogenicity, Safety and Booster Response of Purified Chick Embryo Cell Rabies Vaccine (Pcecv) Administered Intramuscularly or Intradermally to 12- to 18-Month-Old Thai Children Concomitantly With Japanese Encephalitis Vaccine
Brief Title: Rabies Immunization Concomitant With JEV in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Chiron company: Clinical Research and Medical Affairs (Unknown)
Responsible Party: Prof. Arunee Sabchareon, Department of Tropical Pediatrics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M49P2
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-06

CONDITIONS: Rabies
Keywords: rabies vaccination; pre-exposure prophylaxis; rabies virus neutralizing antibody; Antibody response; immunologic memory of rabies vaccination; Safety of rabies vaccination administered in pre-exposure regimens both intramuscular and intradermal routes
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1,2,3,4,5 (Placebo Comparator): 1. Rabies vaccine 1.0 mL IM on day 0, 7, 28,and 1 year
  2. Rabies vaccine 0.5 mL IM on day 0, 7, 28,and 1 year
  3. Rabies vaccine 0.1 mL Intradermal on day 0, 7, 28,and 1 year
  4. Rabies vaccine 0.1 mL Intradermal on day 0, 28,and 1 year
  5. Japanese encephalitis vaccine 0.25 mL subcutaneous
  Interventions: Biological: Rabies vaccine

INTERVENTIONS:
Biological: Rabies vaccine — 1.0 mL IM day 0,7,28 and 1 year

SUMMARY:
Background. The World Health Organization recommends pre-exposure vaccination (PreP) to protect children living in canine rabies endemic countries. Including PreP in national childhood immunization programs (EPI) is a viable option.

Methods. In an open-label phase II clinical trial, 200 healthy toddlers were randomized to receive Purified Chick Embryo Cell Vaccine (PCECV) in a 3-dose Full-IM (1mL), Half-IM (0.5mL), 3-ID (0.1mL), or a 2-dose 2-ID (0.1mL) regimen, all in combination with two doses of Japanese Encephalitis (JEV), or JEV alone. One booster dose of PCECV (IM or ID) and JEV, or JEV alone was administered concomitantly one year after primary vaccination. Safety was evaluated after each injection. Blood was drawn on days 0 and 49, one year later prior to booster and on days 7 and 28 post-booster, and at two and three years post primary vaccination. All sera were analyzed for rabies and JE virus neutralizing antibodies (RVNA, JEVNA).

ELIGIBILITY:
Inclusion Criteria:

* Male and female 12-18 months old toddlers will be included in the study if they;
* are in good health at time of entry into the study as determined by medical history, physical examination and clinical judgment of the investigator;
* are available for all the visits scheduled in the study;
* have been granted a written informed consent signed by their parents

Exclusion Criteria:

* a history of rabies immunization;
* a history of Japanese encephalitis immunization or disease;
* a significant acute or chronic infectious disease at the time of enrollment;
* fever > 38.0 degree C (axillary) or/and significant acute or chronic infection requiring systemic antibiotic or antiviral therapy within the past 7 days before enrollment;
* being under treatment with parenteral, oral and/or inhaled corticosteroids, immunosuppressive drugs or other specific anti-inflammatory drugs or having taken chloroquine during the two months period before enrollment;
* administration of any vaccine within the past 14 days before enrollment;
* known immunodeficiency or an autoimmune disease;
* known hypersensitivity to neomycin, tetracycline, amphotericin-B;
* planned surgery during the study period;
* being enrolled in any other investigational trial contemporaneously;
* the family plans to leave the area of the study site before the end of study period;
* history of febrile convulsions;
* history of wheezing

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2002-08; Primary Completion 2002-10 (Actual); Study Completion 2005-09 (Actual)